CLINICAL TRIAL: NCT05978622
Title: A Multi-country, Post Marketing Observational Study of DME Patients With Suboptimal Response to Anti-VEGF Who Are Initiated With Dexamethasone Intravitreal Implant (DEX-I)
Brief Title: Observational Study of Adult Participants With Diabetic Macular Edema and Suboptimal Response to Anti-Vascular Endothelial Growth Factor Treated With Dexamethasone Intravitreal Implant
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-380
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; DME; Dexamethasone; Dexamethasone Intravitreal Implant; Ozurdex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dexamethasone Intravitreal Implant (DEX-I): Dexamethasone 700 μg intravitreal implant (DEX-I) administered according to general clinical practice.

SUMMARY:
The dexamethasone 700 μg intravitreal implant (DEX-I) delivers dexamethasone gradually to the retina over time. It is an approved drug for the treatment of DME. This study will assess adult participants with diabetic macular edema (DME) and suboptimal response to anti-vascular endothelial growth factor therapy that are treated with DEX-I in the routine clinical setting.

Approximately 327 participants who are prescribed DEX-I by their physicians will be enrolled at approximately 40 sites in approximately 10 countries globally.

Participants will be followed for 18 months post-DEX-I implantation according to the routine clinical practice of the prescribing centers. Only one eye per participant will be evaluated in the study.

No additional burden for participants in this trial is expected.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with DME in the study eye
* Study eye has received at least 3 and no more than 9 anti-VEGF injections in the 12 months prior to DEX-I initiation
* Study eye newly prescribed DEX-I. The prescribing decision lies with the physician and reflects their standard practice
* Participant showing a suboptimal response to anti-VEGF at Baseline in the study eye

Exclusion Criteria:

* Any concomitant ocular or neurologic condition in the study eye that could cause macular edema or affect vision (except cataract)
* History of ocular surgery within 60 days of Baseline in the study eye
* History of Pan-Retinal Photocoagulation (PRP) or sectorial photocoagulation in the study eye in the 3 months prior to Baseline
* Significant media opacities in the study eye limiting Optical Coherence Tomography (OCT) quality
* Uncontrolled Ocular Hypertension (OHT) or advanced glaucoma in the study eye
* Active ocular inflammation in either eye
* Study eyes that are aphakic with Posterior Capsule Rent (PCR), Anterior Chamber Intraocular Lens (ACIOL), iris or scleral-fixed Intraocular Lens (IOL) or history of complicated cataract surgery with PCR
* Prior use of intravitreal corticosteroids in the study eye
* Patients with contraindications to DEX-I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with diabetic macular edema and sub-optimal response to anti-VEGF therapy.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Additional Anti-VEGF Injections after Baseline and before DEX-I Initiation | Baseline to 18 Months
  Number of Additional Anti-VEGF Injections after Baseline and before DEX-I Initiation

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- Belgium (6):
  - Uza /Id# 255831, Edegem, Antwerpen
  - CHU Saint Pierre /ID# 257650, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 255324, Jette, Brussels Capital
  - Ziekenhuis Oost-Limburg /ID# 255934, Genk, Limburg
  - Vitaz /Id# 265553, Sint-Niklaas, Oost-Vlaanderen
  - CHR de la Citadelle /ID# 257254, Liège
- China (5):
  - Shenzhen Eye Hospital /ID# 262954, Shenzhen, Guangdong
  - Tongji Hospital /ID# 270275, Wuhan, Hubei
  - Xi'an Fourth Hospital /ID# 262972, Xi'an, Shaanxi
  - Qingdao Eye Hospital Of Shandong First Medical University /ID# 262756, Qingdao, Shandong
  - West China Hospital, Sichuan University /ID# 262745, Chengdu, Sichuan
- Germany (8):
  - MVZ Augenzentrum am Berliner Ring /ID# 267412, Würzburg, Bavaria
  - MVZ der Klinik Dardenne GmbH Makulazentrum /ID# 269798, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 255660, Leipzig, Saxony
  - Augenzentrum Prinz 25 /ID# 261090, Augsburg
  - Dres. Schubert/Wissmann /ID# 261598, Ettlingen
  - Augenzentrum Frankfurt /ID# 255576, Frankfurt am Main
  - Augenzentrum Frohe Zukunft /ID# 256290, Halle
  - Augenzentrum am Johannisplatz /ID# 255754, Leipzig
- Greece (8):
  - University General Hospital Attikon /ID# 257957, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 258313, Heraklion, Crete
  - University General Hospital of Alexandroupoli /ID# 275850, Alexandroupoli, Evros
  - Eye Clinic of Athens /ID# 258749, Athens
  - General Hospital of Lamia /ID# 265442, Lamia
  - Reg Gen Univ Hosp Larissa /ID# 255235, Larissa
  - Opthalmica SA /ID# 258748, Thessaloniki
  - Papageorgiou General Hospital /ID# 265500, Thessaloniki
- Israel (3):
  - Rabin Medical Center /ID# 265476, Petah Tikva, Central District
  - Kaplan Medical Center /ID# 265471, Rehovot, Central District
  - Tel Aviv Sourasky Medical Center /ID# 265469, Tel Aviv, Tel Aviv
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 258134, Rome, Roma
  - IRCCS Fondazione G.B. Bietti per lo studio e la ricerca in Oftalmologia- ONLUS /ID# 258039, Rome, Roma
  - Universita Politecnica delle Marche - AOU Ospedali Riuniti di Ancona /ID# 258072, Ancona
  - Università di Torino /ID# 258442, Torino
  - ASU FC - P.O. Universitario Santa Maria della Misericordia /ID# 256293, Udine
- Portugal (5):
  - Hospital de Santa Maria Maior, EPE /ID# 261063, Barcelos, Braga District
  - Unidade Local de Saude da Regiao de Leiria, EPE /ID# 262009, Leiria
  - Centro Hospitalar do Baixo Vouga /ID# 264421, Porto
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 262010, Porto
  - Unidade Local de Saude do Estuario do Tejo, EPE /ID# 267945, Vila Franca de Xira
- Taiwan (5):
  - National Taiwan University Hospital /ID# 262426, Taipei City, Taipei
  - Kaohsiung Veterans General Hospital /ID# 262429, Kaohsiung City
  - Far Eastern Memorial Hospital /ID# 262428, New Taipei City
  - China Medical University Hospital /ID# 262427, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 256091, Taoyuan
- United Kingdom (9):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 260908, Plymouth, Devon
  - Gloucestershire Hospitals NHS Foundation Trust /ID# 256886, Cheltenham, Gloucestershire
  - Moorfields Eye Hospital /ID# 258465, London, Greater London
  - Royal Victoria Hospital /Id# 260232, Belfast
  - Bradford Teaching hospitals/ Bradford macular centre /ID# 260909, Bradford
  - Liverpool Univeristy Hospitals NHS Foundation Trust /ID# 260230, Liverpool
  - East Cheshire NHS Trust /ID# 270263, Macclesfield
  - Sunderland Eye Infirmary /ID# 258466, Sunderland
  - Great Western Hospital /ID# 258467, Swindon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-380